CLINICAL TRIAL: NCT03683836
Title: Etiology of Minor Troponin Elevations in Patients With Atrial Fibrillation Visiting Emergency Department
Brief Title: Minor Troponin Elevations in Patients With Atrial Fibrillation
Acronym: Tropo-AF
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, Turku University Hospital
Other Study IDs: T125/2016
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Myocardial Ischemia
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
This study aims at identifying the etiology of troponin-T elevations in patients with atrial fibrillation visiting the emergency department.

DETAILED DESCRIPTION:
The aim of this study is to identify the factors associated with minor cardiac troponin-T elevations in patients presenting in emergency department (ED) with atrial fibrillation (AF) diagnosis , and the possible implications it has on the patients prognosis. Data on 3394 patients from the Turku university hospital catchment area with diagnosis of AF on admission to ED and minor troponin-T elevation were analyzed. Patients were classified into three groups according to the troponin-T value: troponin <15ng/l, 15-50ng/l and 51-100ng/l. Individual patient records were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* two troponin T tests within 72 hours of ED admission
* Prior diagnosis of AF or AF at admission

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation admitted to Turku University Hospital emergency department
Sampling Method: Non-Probability Sample
Enrollment: 3394 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality, myocardial infarction, ischemic stroke | 12 months
  Major adverse cardiac or cerebrovascular event within one year